CLINICAL TRIAL: NCT07159139
Title: Expanded Access Protocol for Vatiquinone in Previously Treated Patients With Inherited Mitochondrial Disease
Brief Title: Vatiquinone Expanded Access Protocol
Acronym: EAP
Status: Available | Type: Expanded Access
Sponsor: Medical University of South Carolina (Other)
Collaborators: PTC Therapeutics (Industry)
Responsible Party: Principal Investigator, Thomas Koch, Professor-Faculty, Medical University of South Carolina
Other Study IDs: Pro00144275
Record Dates: First submitted 2025-06-18; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Mitochondrial Disease
MeSH Terms: conditions — Mitochondrial Diseases | interventions — alpha-tocotrienol quinone

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Vatiquinone — Vatiquinone will be administered per dose and schedule specified in the arm description.

SUMMARY:
The purpose of this study is to provide participants who successfully completed the study titled "An Open-label, Safety Study for Previously Treated Vatiquinone (PTC743) Subjects With Inherited Mitochondrial Disease" with liquid Vatiquinone through an intermediate patient population expanded access protocol.

DETAILED DESCRIPTION:
This expanded access protocol serves to make Vatiquinone accessible to subjects with inherited mitochondrial disease who previously participated in a Vatiquinone clinical trial at the Medical University of South Carolina (MUSC) who in the opinion of the investigator would benefit from continued access to liquid Vatiquinone.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with molecular genetic mitochondrial disease including Leigh syndrome, and Alpers syndrome.
* Completed participation in the study titled "An Open-label, Safety Study for Previously Treated Vatiquinone (PTC743) Subjects With Inherited Mitochondrial Disease"
* In the opinion of the clinical investigator, the continuation to receive Vatiquinone will be of benefit to the participants.
* Enrollment into a clinical trial to receive Vatiquinone is not possible

Exclusion Criteria:

* Current participation in any other interventional study
* Pregnant or currently breast feeding.

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Koch, MD, Principal Investigator — Medical University of South Carolina